CLINICAL TRIAL: NCT03176901
Title: Comparing Mindfulness-Based Stress Reduction With the Health Enhancement Program in the Treatment of Urinary Urge Incontinence in Older Adult Women: A Pilot Feasibility and Randomized Controlled Trial
Brief Title: Comparing Approaches to Treat Older Adult Women's Urge Incontinence: Pilot Feasibility and Randomized Controlled Trial
Acronym: SHUW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Katarina Felsted, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00095461
Record Dates: First submitted 2017-04-27; First posted 2017-06-06 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Urinary Incontinence, Urge; Urinary Incontinence in Old Age
Keywords: urinary urge incontinence; urinary incontinence; older adult women; older adults; mindfulness-based stress reduction; health enhancement program; feasibility; randomized controlled trial; complementary; integrative; therapies
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Two armed study with intervention and comparison groups running parallel to one another
Who Masked: Participant
Masking Description: This is a blinded, randomized controlled trial. Participants are blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): 8 week manualized, standardized mindfulness-based stress reduction program taught by a certified Mindfulness-Based Stress Reduction instructor
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Health Enhancement Program (Active Comparator): 8 week manualized, standardized health enhancement program, taught by a certified health education specialist
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — This experimental arm presents the actual Mindfulness-Based Stress Reduction program as developed in the late seventies and early eighties in its original eight week format
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Health Enhancement Program — This active comparison arm presents the official Health Enhancement Program in its eight week format as developed by MacCoon in 2009.
  Arms: Health Enhancement Program

SUMMARY:
The purpose of this study is to examine the feasibility of conducting a pilot randomized controlled trial comparing mindfulness-based stress reduction with the health enhancement program on symptoms of urinary urge incontinence in older adult women, and to establish preliminary efficacy of these two approaches on symptoms of urinary urge incontinence.

DETAILED DESCRIPTION:
The overarching goal of this research is to evaluate potential treatment options for older women with symptoms of urinary urge incontinence, with a specific focus on Mindfulness-Based Stress Reduction, a promising therapeutic approach in preliminary studies and one increasingly used to treat symptoms associated with brain-visceral interactions. Feasibility and preliminary efficacy will be tested in two randomized study arms: a Mindfulness-Based Stress Reduction intervention group and a Health Enhancement Program intervention comparison group.

This research study will explore the feasibility and preliminary efficacy of treating urinary urge incontinence in older adult women with mindfulness-based stress reduction in comparison to the health enhancement program through a randomized controlled pilot study. Feasibility determinants will include both research feasibility (recruitment, retention, treatment fidelity) and intervention feasibility (acceptability, tolerability, treatment adherence). Clinical outcomes to evaluate preliminary intervention efficacy will include severity of urinary urge incontinence symptoms, bother of urinary urge incontinence symptoms, perceived stress, and perceived level of self-efficacy of self-management of urinary urge incontinence symptoms. Preliminary efficacy of the intervention will also be evaluated with the Patient Global Impression of Improvement, a process measure that rates the patient's "response of a condition to a therapy" (Ryan, n.d., p. 1).

This combined pilot feasibility study and randomized controlled trial will evaluate specific factors crucial to the success of a large trial to evaluate the effect of Mindfulness-Based Stress Reduction on urinary urge incontinence in older adult women. Moore (2011) recommended that the pilot study design parallel the future larger study, particularly when evaluating feasibility in the pilot study. The capacity for hypothesis testing, or establishing causal inference is limited in a pilot study due to insufficient power; however, the information from efficacy testing is vital in informing future larger scale clinical trials. This study will serve as a necessary step for the development of effectiveness trials of Mindfulness-Based Stress Reduction in treatment of urinary urge incontinence in older adult women by informing and guiding evaluation, implementation, and dissemination.

ELIGIBILITY:
Inclusion Criteria:

The following eligibility criteria must be met for the potential participant to be considered for enrollment.

* The study is enrolling older adult women, with urinary urge incontinence.
* They cannot be currently treating their urinary urge incontinence with medication as this will confound results.
* Women who have attempted more extreme treatments and are still experiencing urinary urge incontinence will not be considered as potential participants, as it is unlikely that mindfulness-based stress reduction would treat urinary urge incontinence that is refractory to that degree.
* Participants must be English speaking, as the interventions and homework will be delivered in English.
* postmenopausal women
* Urge predominant urinary incontinence, defined as score of ≥ 3 (moderate to severe urinary incontinence) on the Incontinence Severity Index
* Urge predominant urinary incontinence as determined by question 3 on the 3 Incontinence Questions. The 3 Incontinence Questions has been shown to be a quick and accurate way of diagnosing stress, urge or mixed incontinence in most cases
* Has experienced urinary urge incontinence symptoms for at least three months
* Committed to attend 8 weekly sessions and one half day retreat between weeks 6 and 7
* No pharmacologic therapy for urinary urge incontinence within three weeks of enrollment and no plan to initiate such medications during the 8 week active treatment
* If on hormone therapy or vaginal estrogen, plan to remain on it for the duration of the study; if not on it, no plan to initiate
* No previous intradetrusor Botox injection for urinary urge incontinence and no plan to receive it during the intervention
* No previous neurostimulation for urinary urge incontinence and no plan to receive it during the intervention English speaking
* A score of >24 on the Montreal Cognitive Assessment

Exclusion Criteria:

The following exclusions are applied, as they could seriously limit participation or confound participant response to the intervention:

* Predominantly stress, mixed, or other type of incontinence as determined by question 3 on the 3 Incontinence Questions
* Currently taking medications for Alzheimer's disease or other dementias; these medications could interfere with their participation
* Known neurologic disease acknowledged to impact bladder function including Parkinson's disease, spinal cord injury, or stroke affecting urinary control; these diseases provide cause for urinary urge incontinence and as such the participant would be unlikely to benefit from the intervention
* Current symptomatic urinary tract infection that has not resolved prior to the start of intervention
* Current bladder infection that has not resolved prior to the start of intervention
* Use of an assistive device for ambulation (such as a cane, walker, or wheelchair) and feels that difficulties with bladder management are related to the slowed time in visiting the restroom ("Was urinary urge incontinence a problem before you began using the assistive device?")
* Functionally incontinent, in other words, having a mental or physical condition that prevents a person from visiting the restroom in time
* Ever diagnosed with interstitial cystitis
* Self-report of vaginal bulge protruding outside of the vagina
* Past participation in a formal program of mindfulness-based stress reduction
* Substantial, uncorrected hearing loss
* Substantial, uncorrected vision loss
* Limitations that preclude completing study questionnaires or surveys, such as difficulties with reading and writing or a cognitive impairment

Ages: 55 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — participants must self-identify as female to participate
Enrollment: 25 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Number of potential participants contacted | 10 weeks
  number of people who contacted PI during recruitment process, including the place they heard about the study
number of enrolled participants completing the study | 12 weeks
  number of participants who attended at least five of nine classes number of excused absences number of unexcused absences
percentage of course content delivered during intervention | 44 weeks
  weekly interventionist report on what was taught participants perception of course content delivered measured by a checklist of concepts covered in the weekly interventions at study completion
positive or negative coded responses to the question "How did it go today?" | 8 weeks
  data coded from two participants' responses after each class in each arm
number of participants who completed each week's homework practice | 8 weeks
  participants mark on homework practice log and submit weekly
number of participants recruited for enrollment | 10 weeks
  potential participants who were interested in the study
number of potential participants who are eligible to enroll | 10 weeks
  number of people who passed the screening process via calls or emails
consent rate | 10 weeks
  number of participants who are willing to sign consent document at enrollment interview; number who pass the Montreal Cognitive Assessment and are willing to sign consent document
number of participants enrolled | 10 weeks
  number of people who enrolled into the study
number of dropouts due to stated distress from or dislike of either intervention experience (as opposed to someone needing to withdraw due to a family emergency or illness) | 8 weeks
  participant self-report of what made the intervention challenging - why they were unable or unwilling to complete the course
- number of minutes of homework practice each week | 8 weeks
  totaled from daily numbers reported by participant

SECONDARY OUTCOMES:
change in symptom severity | 16 weeks, 6 months
  measured by the Incontinence Severity Index
change in symptom bother | 16 weeks, 6 months
  measured by the Overactive Bladder questionnaire, short form
change in perceived stress | 16 weeks, 6 months
  measured by the Perceived Stress Scale
change in perceived self-efficacy | 16 weeks, 6 months
  measured by the Geriatric Self Efficacy Index for Urinary Incontinence
self report of rate and trajectory of change in participant impression of improvement | 16 weeks, 6 months
  measured by the Patient Global Impression of Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Katarina F Felsted, MS, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No